CLINICAL TRIAL: NCT05736718
Title: Engaging Clinical Champions to Improve HPV Vaccine Communication and Uptake in Healthcare Systems
Brief Title: Engaging Clinical Champions to Improve HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACTP3CHAMP; 1P01CA250989-01A1 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilloma Virus; vaccination; adolescent medicine; primary care; clinical champions

STUDY DESIGN:
Intervention Model Description: cluster randomized design in which clinics will be randomized within healthcare systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Champion AAT (Experimental): Staff in clinics randomized to this arm will receive an intervention called Announcement Approach Training (AAT). This training is designed to improve communication about HPV vaccination. The training will be organized and delivered by vaccine champions from participating healthcare systems.
  Interventions: Behavioral: Champion Announcement Approach Training
- Traditional AAT (Experimental): Staff in clinics randomized to this arm will also receive Announcement Approach Training (AAT). The training will be organized and delivered by outside experts.
  Interventions: Behavioral: Traditional Announcement Approach Training

INTERVENTIONS:
Behavioral: Champion Announcement Approach Training — AAT is a one-hour communication workshop that trains clinical staff how to recommend HPV vaccine for children ages 9-12. In the champion arm, vaccine champions will deliver the training using slides and a standardized script. They will also conduct outreach and sustainability planning.
  Arms: Champion AAT
Behavioral: Traditional Announcement Approach Training — AAT is a one-hour communication workshop that trains clinical staff how to recommend HPV vaccine for children ages 9-12. In the traditional arm, outside experts will deliver the training using the same slides and script.
  Arms: Traditional AAT

SUMMARY:
This trial will compare two ways to improve communication about HPV vaccination in primary care. The research team will work with primary care clinics. Some clinics will receive communication training from an outside expert. Other clinics will receive the same training from a vaccine champion from their healthcare system.

DETAILED DESCRIPTION:
The researchers will conduct a cluster randomized non-inferiority trial. The trial will compare two ways of delivering a communication workshop called Announcement Approach Training (AAT). AAT is designed to improve communication about HPV vaccination in primary care. The researchers will randomize clinics within participating healthcare systems. Some clinics will receive the training from an outside expert. Other clinics will receive the same training from a vaccine champion from their own system. The researchers will use medical record data to compare changes in HPV vaccination among children ages 9-12. Clinics will be followed for 12 months. The study will engage clinical staff. Researchers will not have direct contact with children or their families.

ELIGIBILITY:
This trial will enroll clinics and intervene with clinical staff. We will use vaccination data from children to evaluate intervention effectiveness. We will not enroll children or interact with them directly.

Inclusion Criteria

Clinics are eligible if they:

* provide primary care to children ages 9-12
* specialize in pediatrics or family medicine

Children's medical records will be eligible to be included in the dataset if children:

* are between the ages of 9-12 years at baseline
* are attributed to a participating clinic at 12-month follow-up

Exclusion criteria

Clinics are excluded if they:

* do not provide primary care to children ages 9-12
* have a specialty other than pediatrics or family medicine

Children's medical records will be excluded if children:

* are not between the ages of 9-12 years at baseline
* are not attributed to a participating clinic at 12-month follow-up
* are receiving hospice/palliative care, are pregnant, or have a history of HPV vaccine contraindications

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who initiate the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline

SECONDARY OUTCOMES:
HPV vaccination (2 doses), 9-12 year olds | from baseline to 12 months
  Proportion of unvaccinated children who complete the HPV vaccine series between baseline and 12-month follow-up, among those who were ages 9-12 at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT05736718/SAP_000.pdf